CLINICAL TRIAL: NCT06990386
Title: Effect of a Self-management Telehealth Program on Improving Strength and Hand Function in Systemic Sclerosis Patients: a Randomized Control Trial
Brief Title: Self-management Telehealth Program for Scleroderma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Orathai Wantha, Registered Nurse, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HE661405; Khon Kaen University (Other: The Research of Khon Kaen University)
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Scleroderma
Keywords: systemic sclerosis; scleroderma and related disorders; exercise; hand function; hand deformity; disability; clinical trials
MeSH Terms: conditions — Scleroderma, Diffuse; Scleroderma, Systemic; Motor Activity; Hand Deformities | interventions — Self-Management

STUDY DESIGN:
Intervention Model Description: An usual education; included booklet that developed based on the self-management framework consisting of 4 categories: a) self-monitoring, which consisted of self-observation and self-recording of DU and RP; b) performing special tasks to manage the disease, including keeping warm, maintaining moisture, and taking traumatic wound precautions; c) information seeking; and d) self-adjustment based on disease activity and treatment Video guide ; was the hand and joint exercise video guide that included a 3.27-minute educational video on 6 basic daily hand exercises including: a) stretching wrist flexion and extension, b) range of motion (ROM) ulnar and radial deviation, c) ROM finger abduction and adduction, d) finger pincer, e) finger flexion and extension, and f) finger grab Telephone notifications ; consisted of weekly calls for further continuity and engagement with hand exercises. Each call lasted about 10 minutes, providing problem-solving support, knowledge reinforcement
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- usual education (Other): An usual education included self-management booklet that developed based on the self-management framework consisting of 4 categories: a) self-monitoring, which consisted of self-observation and self-recording of DU and RP; b) performing special tasks to manage the disease, including keeping warm, maintaining moisture, and taking traumatic wound precautions; c) information seeking; and d) self-adjustment based on disease activity and treatment.
  Interventions: Behavioral: self-management program
- Video guide and usual education (Active Comparator): Video guide add on usual education was the hand and joint exercise video guide that included a 3.27-minute educational video on 6 basic daily hand exercises including: a) stretching wrist flexion and extension, b) range of motion (ROM) ulnar and radial deviation, c) ROM finger abduction and adduction, d) finger pincer, e) finger flexion and extension, and f) finger grab.
  Interventions: Behavioral: Video guide and usual education
- Telephone notification, video guide and usual education (Active Comparator): Telephone notifications consisted of weekly calls for further continuity and engagement with hand exercises. Each call lasted about 10 minutes, providing problem-solving support, knowledge reinforcement, and motivation to encourage adherence to the program.
  Interventions: Behavioral: Telephone notification, video guide and usual education

INTERVENTIONS:
Behavioral: self-management program — Self-management booklet based on the self-management framework consisting of 4 categories: a) self-monitoring, which consisted of self-observation and self-recording of DU and RP; b) performing special tasks to manage the disease, including keeping warm, maintaining moisture, and taking traumatic wound precautions; c) information seeking; and d) self-adjustment based on disease activity and treatment.
  Arms: usual education
Behavioral: Video guide and usual education — Video guide was the hand and joint exercise video guide that included a 3.27-minute educational video on 6 basic daily hand exercises including: a) stretching wrist flexion and extension, b) range of motion (ROM) ulnar and radial deviation, c) ROM finger abduction and adduction, d) finger pincer, e) finger flexion and extension, and f) finger grab.
  Arms: Video guide and usual education
Behavioral: Telephone notification, video guide and usual education — Telephone notifications consisted of weekly calls for further continuity and engagement with hand exercises. Each call lasted about 10 minutes, providing problem-solving support, knowledge reinforcement, and motivation to encourage adherence to the program.
  Arms: Telephone notification, video guide and usual education

SUMMARY:
Scleroderma causes the skin on the hands to harden, causing the hands to contract, and the fingers to bend abnormally, which affect the patient's work and quality of life.

This project aims to test the effect of a self-management telehealth program. The goal of this clinical trial is to improving hand strength and function in SSc patients.

Participants will: randomly into 3 groups; a) usual education, b) watching 3.27-minute video guide as needed adding on usual education, c) watching video guide and weekly telephone notifications adding to usual education.

A physical therapist coached home program for self-hand and joint exercise, a nursing coach home routine hand care.

Visit the clinic with a diary at 6 weeks after program for checkups and tests

Researchers will compare hand strength and function, self-management behavior, HAMIS scores, hand grip strength (HGS), and quality of life (QoL) between groups, as well as the changes in these parameters at week 6 compared to baseline.

ELIGIBILITY:
Inclusion Criteria:

Adult SSc patients who met the 2013 classification criteria of the American College of Rheumatology/European Alliance of Associations for Rheumatology and fulfilled all of the following criteria were included:

* Ability to communicate in the Thai language
* Stable disease
* Hand involvement defined as a hand mobility in scleroderma score ≥1 or a limited range of motion in at least one hand joint
* Ownership of a smartphone capable of recording video clips
* Ability to access videos on their smartphone independently

Exclusion Criteria:

* Severe contracture deformity of the hands (defined as a hand mobility in scleroderma score of 27)
* Impaired hand sensation; cognitive, hearing, or visual impairment; or physical limitations (e.g., paralysis, muscle weakness)
* Scheduled surgery involving the hand, eyes, or ears; or required hospitalization within the past 6 weeks
* Presence of infected wounds or active inflammation on the hand, wrist, or fingers that prevents performance of hand exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-08-29 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Hand grip strength | 6 weeks

SECONDARY OUTCOMES:
Hand mobility in scleroderma score | 6 weeks
  The hand mobility in scleroderma score includes 9 items that assess finger flexion and extension, thumb abduction, pincer grip, finger adduction, volar flexion of the wrist, dorsal extension, and pronation and supination of the forearm. Each item is scored from 0 (fully performed) to 3 (unable to perform). The total score ranged from 0 to 27, with higher scores indicating worse hand mobility.
Visual analog scale of Quality of life | 6 weeks
  The health status quality of life self-assessment is assessed via a visual analog scale from 0 to 100.
Self-management behavior score | 6 weeks
  The Self-Management Behavior Questionnaire consisted of an 11-item questionnaire using a 4-point Likert scale (1 = never, 4 = always) to assess patients based on the self-management framework. The total score ranged from 11 to 44. A higher score indicated better self-management behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No